CLINICAL TRIAL: NCT00249925
Title: Enhancing Function of Frail Elders At Home
Brief Title: Project ABLE:Advancing Better Living for Elders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: R01AG013687 (NIH)
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Frail Elderly
Keywords: Home modification; Occupational Therapy; Physical Therapy; Home care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Home-Based Intervention
Behavioral: Multi-component home-based intervention

SUMMARY:
The specific aims of the study are to: 1) test the effectiveness of a home-bases intervention to improve home safety, fall efficacy and functional performance; 2) determine if the use of environmental strategies results in occurrence of less negative health events (falls and depression); 3) compare types of environmental strategies accepted and used under different treatment conditions; and 4) evaluate the cost-effectiveness of the intervention program.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* community dwelling
* functional vulnerability/HRCA vulnerability index= >1 problem area

Exclusion Criteria:

* Mini-Mental Status Examination (MMSE) score of less than or equal to 23
* legal blindness
* bed bound
* nursing home placement or relocation expected within 12 months of study eligibility

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 319
Dates: Start 2000-01; Primary Completion 2004-06 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Functional difficulty
Fear of falling
Self-efficacy

SECONDARY OUTCOMES:
Home hazards
Control oriented strategy use
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Laura N Gitlin, Ph.D, Principal Investigator — Thomas Jefferson University
Locations (1):
- Philadelphia Corporation for Aging (PCA), Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Rose KC, Gitlin LN, Dennis MP. Readiness to use compensatory strategies among older adults with functional difficulties. Int Psychogeriatr. 2010 Dec;22(8):1225-39. doi: 10.1017/S1041610210001584. Epub 2010 Jul 27. PMID 20663239